CLINICAL TRIAL: NCT03147352
Title: ProTreat - Prognosis and Treatment of Necrotizing Soft Tissue Infections: A Prospective Cohort Study
Brief Title: Prognosis and Treatment of Necrotizing Soft Tissue Infections: A Prospective Cohort Study
Acronym: ProTreat
Status: Completed | Type: Observational
Sponsor: Ole Hyldegaard (Other)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor-Investigator, Ole Hyldegaard, Clinical Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: PROTREAT1-PP-2017
Record Dates: First submitted 2017-04-26; First posted 2017-05-10 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Necrotizing Soft Tissue Infection; Necrotizing Fascitis; Gas Gangrene; Fournier Gangrene
Keywords: Fasciitis; Gangrene; Fasciitis, Necrotizing; Soft Tissue Infections; Fournier's Gangrene; Streptococcal septic shock syndrome; Flesh eating bacteria; Meleneys ulcer; Wounds and Injuries; Streptococcus pyogenes; Staphylococcus aureus; Soft Tissue Infections/blood; Necrosis/blood; Necrosis/diagnosis; Necrosis/mortality; Necrosis/surgery; Prognosis; Risk Factors; Bacterial Infections; Infection; Skin Diseases, Bacterial; Observational study; Biological markers; Endothelium; suPAR; sTM; syndecan-1; sE-selectin; VE-cadherin; protein C; Hyperbaric oxygen therapy; HBOT
MeSH Terms: conditions — Fasciitis, Necrotizing; Gas Gangrene; Fournier Gangrene; Fasciitis; Gangrene; Soft Tissue Infections; Wounds and Injuries; Staphylococcal Infections; Necrosis; Disease; Bacterial Infections; Infections; Skin Diseases, Bacterial | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Whole blood and plasma/serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSTI patients: NSTI is an infection that requires acute hospitalization with intensive care treatment and/or surgery as a consequence of severe soft tissue infection in subcutis, muscle and/or fascia and that spreads along tissue structures.
  Interventions: Device: Hyperbaric oxygen therapy
- Orthopaedic control patients: Elective orthopaedic control patients.

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy with 100 % oxygen at 1.8 ATA for 2 hours.
  Groups: NSTI patients

SUMMARY:
The investigators will analyze biomarkers related to the prognosis and treatment of necrotizing soft tissue infections (NSTI). The focus will be on whether certain endothelial and immune system biomarkers can function as markers of disease severity, mortality as well as the effects of hyperbaric oxygen therapy (HBOT). Biomarkers will be measured upon admission to an intensive care unit at Copenhagen University Hospital and during the following 3 days.

DETAILED DESCRIPTION:
Introduction:

Necrotizing soft-tissue infections (NSTI) are among the most serious and deadly infections known. They are characterized by rapidly progressing soft-tissue inflammation with necrosis and can quickly cause multiple organ failure and death. Mortality has been shown to be 25-35 %, with survivors coping with amputations and prolonged rehabilitation.

Currently, there is a lack of proper tools to evaluate the severity and prognosis of NSTI in individual patients. This results in necessary, yet sometimes overzealous surgical debridement, culminating in prolonged patient rehabilitation and invalidity. Hyperbaric oxygen therapy (HBOT) may be added as adjunctive therapy of NSTI. However, there is no clear understanding of the effectiveness of HBOT on NSTI. The investigators seek to remedy these two issues by examining multiple biomarkers over the course of several studies.

Methodology:

Location: Copenhagen University Hospital, Rigshospitalet, Denmark.

Design: Observational cohort study.

Cohort: All NSTI patients in Denmark since 2013.

Controls: 50-100 Patients undergoing elective, orthopedic surgery at Rigshospitalet.

Biomarkers: soluble thrombomodulin, syndecan-1, sE-selectin, VE-cadherin, protein C, suPAR.

Sample size calculations:

1: The test kits the investigators will be using to measure the primary outcome sTM (Human sCD141 ELISA kit, Nordic Biosite) have an interassay standard variation of 0.58 ng/ml. In order to be certain that measured changes in sTM concentration are not a result of interassay standard deviation, the investigators have set the mimimum relevant difference in sTM to 3 x the interassay standard variation, thus 1.75 ng/ml.

The investigators prepared a power calculation using a Wilcoxon rank sum test. Assuming an estimated standard deviation of 4.6 ng/ml and a mean of 9.9 ng/ml, the investigators will need to include a maximum of 150 NSTI patients and 50 elective surgery patients to reach a statistical power of at the very least 60 % (a very conservative estimate) and presumably closer to 85 % (more realistic estimate) at a 5 % significance level. The estimates depend on data distribution.

2: The test kits the investigators will be using to measure the primary outcome sE-selectin (Human CD62E ELISA kit, Diaclone) have an interassay standard variation of 0.37 ng/ml. In order to be certain that measured changes in sE-selectin concentration are not a result of interassay standard variation, the investigators have set the mimimum relevant difference in sE-selectin to 3 x the interassay standard variation, thus 1.1 ng/ml.

Assuming an estimated standard deviation of 209 ng/ml (septic shock) vs. 23 ng/ml (severe sepsis and sepsis) and means of 295 vs. 181 ng/ml, respectively, the investigators will need to include at least 132 NSTI patients and 50 elective surgery patients to reach a statistical power of 90 % at a 5 % significance level.

3: suPAR levels during NSTI have never previously been examined. In order to estimate sample size and since NSTI patients are also septic, the investigators are basing the sample size calculation on a previous study concerning the correlation between suPAR and sepsis. This study found statistically significant correlation between suPAR levels and mortality in 141 patients. This is also the goal of this study. Further studies have also found significant correlations between suPAR, sepsis and mortality in 132 patients. The investigators will include at least 150 NSTI patients during this study.

Statistical considerations:

To check whether the HBOT treatment has an effect on the range of biomarkers, the investigators will analyze the means and variances of the biomarkers in the NSTI group and the two control groups, the orthopaedic patients and the sepsis patients. Non-parametric data will be log-transformed and will be presented as median values with IQR. Wilcoxon rank sum tests will be used for group comparisons. Fisher's exact test will be used for categorical data. Correlation analysis will be performed using Spearman rank correlation or Pearson correlation. To assess the quality of suPAR as a predictor of health outcomes, a model selection exercise will be conducted with various types of regression models. The type of regression will vary with the type of health-outcome, with suPAR as the predictor in all cases. Receiver operating characteristic (ROC) curve analysis will be applied to determine suPARs accuracy as a marker of severity and mortality in patients with NSTI. The investigators will construct Kaplan-Meier curves for survival data. Statistically significant results are when p<0.05.

Data:

Data will be handled according to the National Data Protection Agency. All original records (including consent forms and questionnaires) will be archived at the trial site for 15 years. The National Data Protection Agency has approved the biobank (RH-2016- 199). Data checks have been programmed into the data registry to warn when input variables are outside of predefined possible clinical range. All registry data will be compared to external data sources, i.e. medical records, to ensure accuracy. Standard Operating Procedures have been implemented regarding data collection. Patients with missing data for calculating for example SAPS II scores etc. will be excluded from the study.

Ethics:

The trial will adhere to the Helsinki Declaration and Danish law. The National Ethics Committee and the Regional Ethics Committee (H-16021845) have approved this study.

Biomarker analyses, data extraction and interpretation will be performed once the recruitment of participants has ended.

ELIGIBILITY:
Inclusion criteria for NSTI patients (both of which must be met):

* Diagnosed with NSTI based on surgical findings (necrosis of any soft tissue compartment; dermis, hypodermis, fascia or muscle)
* Admitted to the Intensive Care Unit (ICU) and/or operated for NSTI at Copenhagen University Hospital

Exclusion Criteria for NSTI patients:

* They are categorized as non NSTI in the operating theatre

Inclusion criteria for orthopaedic control patients:

* Undergoing elective orthopedic surgery (non-pathological fractures, joint replacement surgery or spine surgery) at Copenhagen University Hospital

Exclusion criteria for orthopaedic control patients:

* Ongoing infection or inflammatory condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSTI cohort:
  All NSTI patients treated at the University Hospital of Copenhagen, Rigshospitalet.
  Orthopaedic control cohort:
  Undergoing elective orthopedic surgery (non-pathological fractures, joint replacement surgery or spine surgery) at Copenhagen University Hospital
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
sTM and sE-selectin as biomarkers of HBOT effect in NSTI patients | At admission, and during the next 3 days in the ICU
  Changes in plasma sTM and sE-selectin concentrations in NSTI patients, compared with the control group
suPAR as a biomarker of disease severity and prognosis in NSTI patients with and without septic shock | At admission
  Association between plasma suPAR levels and NSTI mortality, and SAPS II and SOFA scores

SECONDARY OUTCOMES:
Mortality | While in the ICU, and at 28, 90, 180 days
  Mortality
Amputation rate | During ICU admission (expected average of 8 days)
  At any anatomical site
ICU scoring systems | During ICU admission (expected average of 8 days)
  SAPS II (day 1) APACHE II (day 1) SOFA, GCS excluded (day 1-7)
Multiple organ failure | During ICU admission (expected average of 8 days)
  Multiple organ failure
Debridements | During ICU admission (expected average of 8 days)
  Number of debridements
Microbial etiology | During ICU admission (expected average of 8 days)
  Tissue and blood samples
Time from admission to primary hospital until first surgery/debridement | 2 days
Ventilator treatment | During ICU admission (expected average of 8 days)
  Ventilator treatment during stay at ICU
Renal replacement therapy | During ICU admission (expected average of 8 days)
  Renal replacement therapy during stay at ICU
Vasopressor treatment | During ICU admission (expected average of 8 days)
  Vasopressor treatment during stay at ICU
Steroid treatment | Up to 7 days before surgical diagnose at primary hospital
  Steroid treatment (injection/oral intake) up to development of NSTI
HBOT and endothelial biomarkers | At admission, and the next 3 days in the ICU
  Any differences in sTM, syndecan-1, sE-selectin, VE-cadherin and protein C levels between NSTI patients who do not receive HBOT within the first 24 hours of ICU admission (because they are deemed too unstable for HBOT) vs. those who receive HBOT within the first 12 and 24 hours of ICU admission
Biomarkers and disease severity | At admission, and the next 3 days in the ICU
  Systemic inflammatory response syndrome, sepsis, severe sepsis and septic shock will be diagnosed according to standardized criteria (American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference Committee) and suPAR, sTM and sE-selectin will be investigated to see if there is a correlation between disease severity in these groups

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Polzik, MD, Principal Investigator — Rigshospitalet, Denmark; Ole Hyldegaard, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kayal S, Jais JP, Aguini N, Chaudiere J, Labrousse J. Elevated circulating E-selectin, intercellular adhesion molecule 1, and von Willebrand factor in patients with severe infection. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):776-84. doi: 10.1164/ajrccm.157.3.9705034. PMID 9517590
- [Background] Huttunen R, Syrjanen J, Vuento R, Hurme M, Huhtala H, Laine J, Pessi T, Aittoniemi J. Plasma level of soluble urokinase-type plasminogen activator receptor as a predictor of disease severity and case fatality in patients with bacteraemia: a prospective cohort study. J Intern Med. 2011 Jul;270(1):32-40. doi: 10.1111/j.1365-2796.2011.02363.x. Epub 2011 Mar 21. PMID 21332843
- [Background] Backes Y, van der Sluijs KF, Mackie DP, Tacke F, Koch A, Tenhunen JJ, Schultz MJ. Usefulness of suPAR as a biological marker in patients with systemic inflammation or infection: a systematic review. Intensive Care Med. 2012 Sep;38(9):1418-28. doi: 10.1007/s00134-012-2613-1. Epub 2012 Jun 16. PMID 22706919
- [Background] Blann A, Seigneur M. Soluble markers of endothelial cell function. Clin Hemorheol Microcirc. 1997 Jan-Feb;17(1):3-11. PMID 9181753
- [Background] Buras JA, Stahl GL, Svoboda KK, Reenstra WR. Hyperbaric oxygen downregulates ICAM-1 expression induced by hypoxia and hypoglycemia: the role of NOS. Am J Physiol Cell Physiol. 2000 Feb;278(2):C292-302. doi: 10.1152/ajpcell.2000.278.2.C292. PMID 10666024
- [Background] Reitsma S, Slaaf DW, Vink H, van Zandvoort MA, oude Egbrink MG. The endothelial glycocalyx: composition, functions, and visualization. Pflugers Arch. 2007 Jun;454(3):345-59. doi: 10.1007/s00424-007-0212-8. Epub 2007 Jan 26. PMID 17256154
- [Background] Rehm M, Bruegger D, Christ F, Conzen P, Thiel M, Jacob M, Chappell D, Stoeckelhuber M, Welsch U, Reichart B, Peter K, Becker BF. Shedding of the endothelial glycocalyx in patients undergoing major vascular surgery with global and regional ischemia. Circulation. 2007 Oct 23;116(17):1896-906. doi: 10.1161/CIRCULATIONAHA.106.684852. Epub 2007 Oct 8. PMID 17923576
- [Derived] Polzik P, Johansson PI, Hyldegaard O. How biomarkers reflect the prognosis and treatment of necrotising soft tissue infections and the effects of hyperbaric oxygen therapy: the protocol of the prospective cohort PROTREAT study conducted at a tertiary hospital in Copenhagen, Denmark. BMJ Open. 2017 Oct 5;7(10):e017805. doi: 10.1136/bmjopen-2017-017805. PMID 28982834